CLINICAL TRIAL: NCT01413659
Title: Evaluation of the Effect of Preoperative Symbiotic Bowel Conditioning on Surgical Site Infection After Elective Colorectal Surgery
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: HamidReza Naderi, Imam Reza General Hospital - Surgical Oncology Research Center (SORC)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MUMS-89619
Record Dates: First submitted 2011-08-08; First posted 2011-08-10 (Estimated); Last update posted 2011-08-25 (Estimated); Status verified 2011-07

CONDITIONS: Postoperative Wound Infection
Keywords: Colorectal surgery; Surgical site infection; Symbiotic
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (1):
- Symbiotic (Experimental): Symbiotic is a combination of prebiotics and probiotics that is designed to have synergistic or additive effects benefiting the host
  Interventions: Biological: Symbiotic

INTERVENTIONS:
Biological: Symbiotic — Oral symbiotic every 8 h since 2 days before operation; Symbiotic resumes postoperatively on day +2 until day +4 for a total of 4 d of treatment (12 doses).

SUMMARY:
The objective of the study is to investigate whether peri-operative symbiotic treatment could reduce the risk of postoperative infections in patients undergoing elective colorectal surgery. This study was also designed to assess the risk-adjusted incidence and predictors of surgical site infections.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders
2. More than 14 years old
3. Candidate for elective colorectal surgery

Exclusion Criteria:

1. Denied written informed consent,
2. Severe neutropenia, and
3. Critically ill condition
4. Not meeting inclusion criteria

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-12 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Frequency of post-operative infection after elective colorectal surgery among patients with and without pre-operative symbiotic conditioning. | 15 months

SECONDARY OUTCOMES:
The incidence of postoperative infection including surgical site infections (SSIs) and distant-site infections after elective colorectal surgery in patients whether or not receiving pre-operative symbiotic conditioning. | 15 months